CLINICAL TRIAL: NCT01461980
Title: A Phase 2, Randomized, Active-controlled, Observer-blinded Trial, To Assess The Safety, Tolerability, And Immunogenicity Of Mcv4, Tdap Vaccine And Bivalent Rlp2086 Vaccine When Administered Concomitantly In Healthy Subjects Aged > = 10 To <13 Years
Brief Title: A Clinical Trial to Study the Safety, Tolerance and Immunogenic Response to MCV4, Tdap and Bivalent rLP2086 Vaccine When Given at the Same Time to Children Between the Ages of 10 Through 12 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Quadruple | Purpose: Prevention
Other Study IDs: B1971015; 6108A1-2005 (Other: Alias Study Number)
Record Dates: First submitted 2011-09-28; First posted 2011-10-28 (Estimated); Results first posted 2015-05-25 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-11

CONDITIONS: Vaccines; Meningococcal Vaccines
Keywords: vaccine; rLP2086; MCV4; Tdap; meningitis B; N. meningitidis serogroup B; adolescents; observer-blind
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MCV4 + Tdap+ rLP2086 (Active Comparator): Group 1 - MCV4 + Tdap + rLP2086
  Interventions: Biological: rLP2086 + MCV4 + Tdap
- MCV4 + Tdap + saline (Active Comparator): Group 2, MCV4 + Tdap+ saline
  Interventions: Biological: MCV4 + Tdap + saline
- Saline + saline + rLP2086 (Placebo Comparator): Group 3- rLP2086 + saline
  Interventions: Biological: rLP2086 + saline

INTERVENTIONS:
Biological: rLP2086 + MCV4 + Tdap — At visit 1, group 1 will receive MCV4 + Tdap vaccines concomitantly with an injection of rLP2086. At visits 3 and 5 (Months 2 and 6), group 1 will receive an injection of rLP2086.
  Arms: MCV4 + Tdap+ rLP2086
Biological: MCV4 + Tdap + saline — At visit 1, group 2 will receive MCV4 + Tdap vaccines concomitantly with an injection of saline. At visits 3 and 5 (months 2 and 6), this group will receive a saline injection only.
  Arms: MCV4 + Tdap + saline
Biological: rLP2086 + saline — At visit 1, group 3 will receive 2 injections of saline concomitantly with an injection of rLP2086. At visits 3 and 5 (Months 2 and 6), group 3 will receive an injection of rLP2086. Subjects randomized to this group will receive MCV4 and Tdap following their final visit blood draw (Visit 6).
  Arms: Saline + saline + rLP2086

SUMMARY:
This is a clinical study to assess the safety, tolerance and immunogenic response to MCV4(quadrivalent meningococcal polysaccharide conjugate, meningococcal serogroups A,C,Y, and W135), Tdap (diphtheria, tetanus, and acellular pertussis), and bivalent rLP2086 vaccine. Healthy male and female subjects, between the ages of 10 to 12 years old, will be randomized into 1 of 3 groups. The subjects, investigators, site staff and sponsor will be blinded to all injections given throughout the study. An unblinded administrator will be responsible to administer the vaccinations to all subjects and will be unblinded to the subject randomization in order to determine which subjects were in randomized to group 3 so they may receive their catch-up vaccinations of MCV4 and Tdap. A final telephone contact will be conducted with all subjects 6-months post their last vaccination to obtain safety information.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject (and a legally authorized representative) has been informed of all pertinent aspects of the study.
* Parent /legally authorized representative and subjects who are willing and able to comply with scheduled visits, laboratory tests, and other study procedures.
* Male or female subject aged greater than or equal to 10 and <13 years at the time of enrollment.
* Available for the entire study period and can be reached by telephone.
* Healthy subject as determined by medical history, physical examination, and judgment of the investigator.
* Has received full series (5-dose series is preferred, 4-dose catch up series is allowed) of diphtheria, tetanus and pertussis (whole cell or acellular) vaccines per country specific recommendations applicable at the time of receipt.
* Male and female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study.

Exclusion Criteria:

* Previous vaccination with any meningococcal serogroup B vaccine.
* Vaccination with any diphtheria, tetanus or pertussis vaccine within 5 years of the first study vaccination.
* Previous vaccination with any MCV4 vaccine.
* A previous anaphylactic reaction to any vaccine or vaccine-related component.
* Contraindication to vaccination with MCV4 and/or Tdap vaccine.
* Subjects receiving any allergen immunotherapy with a non-licensed product or receiving allergen immunotherapy with a licensed product and are not on stable maintenance doses.
* Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection.
* A known or suspected defect of the immune system that would prevent an immune response to the vaccine, such as subjects with congenital or acquired defects in B cell function, those receiving chronic systemic (oral, intravenous or intramuscular) corticosteroid therapy, or those receiving immunosuppressive therapy. Subjects with terminal complement deficiency may not be included.
* History of culture-proven disease caused by Neisseria meningitidis or Neisseria gonorrhoea.
* Significant neurological disorder or history of seizure (excluding simple febrile seizure).
* Receipt of any blood products, including immunoglobulin within 6 months before the first study vaccination.
* Current chronic use of systemic antibiotics.
* Any neuroinflammatory or autoimmune condition, including, but not limited to, transverse myelitis, uveitis, optic neuritis, and multiple sclerosis.

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2648 (Actual)
Dates: Start 2011-09-28 (Actual); Primary Completion 2014-05-08 (Actual); Study Completion 2014-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (113):
- United States (113):
  - Radiant Research, Inc., Birmingham, Alabama
  - Costal Clinical Research, Inc., Daphne, Alabama
  - Clinical Research Advantage Inc/ East Valley Family Physicians, PLC, Chandler, Arizona
  - Radiant Research, Inc., Chandler, Arizona
  - Clinical Research Advantage, Inc./Mesa Family Medical Center, PC, Mesa, Arizona
  - Clinical Research Advantage, Inc./Desert, Mesa, Arizona
  - Radiant Research, Inc., Tucson, Arizona
  - The Children's Clinic of Jonesboro, PA, Jonesboro, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - Kaiser Permanente Fresno, Fresno, California
  - Kaiser Permanente Hayward, Hayward, California
  - Pediatric Care Medical Group, Huntington Beach, California
  - Loma Linda University, Loma Linda, California
  - Loma Linda University Health Care Pediatric Clinic, Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Loma Linda University Health Care - Moreno Valley Pediatrics, Moreno Valley, California
  - Bayview Research Group, LLC, Paramount, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Kaiser Permanente Sacramento, Sacramento, California
  - California Research Foundation, San Diego, California
  - Bayview Research Group, LLC, Valley Village, California
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Colorado Springs Family Practice, Colorado Springs, Colorado
  - Radiant Research, Inc., Denver, Colorado
  - Norwich Pediatric Group, P.C., Norwich, Connecticut
  - University of South Florida, Tampa, Florida
  - Emory University School of Medicine Department of Pediatrics, Atlanta, Georgia
  - Emory University School of Medicine, Atlanta, Georgia
  - Radiant Research, Inc, Atlanta, Georgia
  - North Georgia Clinical Research Center dba Whites Pediatrics, Dalton, Georgia
  - Pediatrics and Adolescent Medicine, PA, Marietta, Georgia
  - Pediatrics and Adolescent Medicine, Woodstock, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Northern Illinois Research Associates, DeKalb, Illinois
  - Clinical Research Advantage, Inc./ Ridge Family Practice, PC, Council Bluffs, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Via Christi Clinic, P.A., Wichita, Kansas
  - Kentucky Pediatric/Adult Research, Bardstown, Kentucky
  - University of Louisville Pediatrics: Children and Youth Project, Louisville, Kentucky
  - Brownsboro Park Pediatrics, Louisville, Kentucky
  - Bluegrass Clinical Research, Inc., Louisville, Kentucky
  - Southwestern Medical Clinic Lakeland Healthcare Affiliate, Stevensville, Michigan
  - Allina Health Bandana Square Clinic, Saint Paul, Minnesota
  - Aspen Medical Group/ Odyssey Research, Saint Paul, Minnesota
  - Aspen Medical Group, Saint Paul, Minnesota
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Radiant Research, Inc., St Louis, Missouri
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Clinical Research Advantage, Inc. / Prairie Fields Family Medicine, PC, Fremont, Nebraska
  - Midwest Children's Health Research Institute, Lincoln, Nebraska
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - Creighton Pediatric Infectious Diseases Creighton University Medical Center, Omaha, Nebraska
  - Clinical Research Center of Nevada, Henderson, Nevada
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Child Health Care Associates, East Syracuse, New York
  - Duke University Medical Center - Duke Health Center, Durham, North Carolina
  - Durham Pediatrics, Durham, North Carolina
  - Duke Health Center, Durham, North Carolina
  - PMG Research of Raleigh, LLC -, Raleigh, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - Innovis Health, Fargo, North Dakota
  - Odyssey Research, Fargo, North Dakota
  - Radiant Research, Inc, Akron, Ohio
  - Cincinnati Center for Clinical Research, Satellite Site - Clinic, Cincinnati, Ohio
  - Cincinnati Childrens Hospital Medical Center Gamble Program for Clinical Studies, Cincinnati, Ohio
  - Dr. Shelly David Senders, MD Inc. dba Senders Pediatrics, Cleveland, Ohio
  - Senders Pediatrics, Cleveland, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Radiant Research, Columbus, Ohio
  - Ohio Pediatric Research Association, Dayton, Ohio
  - Ohio Pediatrics, Inc., Dayton, Ohio
  - Ohio Pediatrics, Inc., Huber Heights, Ohio
  - Ohio Pediatric Research, Kettering, Ohio
  - Christopher Brad Redden, ARNP Healthcare One Urgent Care and Family Practice, El Reno, Oklahoma
  - Lynn Institute of Norman (LION), Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma State University - Center for Health Sciences - Pediatric Research, Tulsa, Oklahoma
  - Office of Richard Ohnmacht, Cranston, Rhode Island
  - Omega Medical Research, Warwick, Rhode Island
  - Radiant Research, Inc., Anderson, South Carolina
  - Charleston Pediatrics, Charleston, South Carolina
  - PMG Research of Charleson, Mt. Pleasant, South Carolina
  - Internal Medicine & Pediatric Associates of Bristol, PC, Bristol, Tennessee
  - PMG Research of Bristol, Bristol, Tennessee
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - Tekton Research, Inc., Austin, Texas
  - Radiant Research, Inc., Dallas, Texas
  - Advances in Health Research, Inc, Houston, Texas
  - West Houston Clinical Research Service, Houston, Texas
  - Pediatric Healthcare of Northwest Houston, Houston, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Child Care Associates, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Radiant Research, Inc., San Antonio, Texas
  - First Steps Pediatrics, San Antonio, Texas
  - Pediatric Healthcare of Northwest Houston, PA, Tomball, Texas
  - Pediatric Healthcare of Northwest Houston, Tomball, Texas
  - Radiant Research, Inc., Murray, Utah
  - J. Lewis Resarch Incorporated, Foothill Family Clinic, Salt Lake City, Utah
  - J. Lewis Research Inc. - Foothill Family Clinic South, Salt Lake City, Utah
  - Jean Brown Research, Salt Lake City, Utah
  - J. Lewis Research, Inc. - Jordan River Family Medicine, South Jordan, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - PI-Coor Clinical Research, LLC, Burke, Virginia
  - Pediatric Associates of Charlottesville, PLC, Charlottesville, Virginia
  - Pediatric Associates of Charlottesville, PLC - West Satellite, Charlottesville, Virginia
  - Pediatric Associates of Charlottesville, PLC - North Satellite, Charlottesville, Virginia
  - The Vancouver Clinic, Vancouver, Washington
  - Gundersen Clinic, LTD, La Crosse, Wisconsin
  - Monroe Clinic, Monroe, Wisconsin

REFERENCES:
- [Derived] Beeslaar J, Mather S, Absalon J, Eiden JJ, York LJ, Crowther G, Maansson R, Maguire JD, Peyrani P, Perez JL. Safety data from the MenB-FHbp clinical development program in healthy individuals aged 10 years and older. Vaccine. 2022 Mar 15;40(12):1872-1878. doi: 10.1016/j.vaccine.2022.01.046. Epub 2022 Feb 11. PMID 35164991
- [Derived] Beeslaar J, Peyrani P, Absalon J, Maguire J, Eiden J, Balmer P, Maansson R, Perez JL. Sex, Age, and Race Effects on Immunogenicity of MenB-FHbp, A Bivalent Meningococcal B Vaccine: Pooled Evaluation of Clinical Trial Data. Infect Dis Ther. 2020 Sep;9(3):625-639. doi: 10.1007/s40121-020-00322-5. Epub 2020 Jul 17. PMID 32681472

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 2648 participants were enrolled in this study. Of these, 19 participants were randomized but did not receive study vaccination.
Groups:
- MCV4+Tdap+rLP2086: Randomized to receive Quadrivalent meningococcal polysaccharide conjugate (MCV4) and Tetanus, diphtheria, and acellular pertussis (Tdap) vaccine on 0- month, Neisseria meningitidis serogroup B (MnB) bivalent recombinant lipoprotein 2086 (rLP2086) vaccine on a 0-, 2-, 6- month schedule.
- MCV4+Tdap+Saline: Randomized to receive MCV4 and Tdap vaccine on 0- month, Saline on a 0-, 2-, 6- month schedule.
- Saline+Saline+rLP2086: Randomized to receive Saline on 0- month, rLP2086 vaccine on a 0-, 2-, 6- month schedule, MCV4 and Tdap vaccine on 7- month.
Period: Overall Study
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline | Saline+Saline+rLP2086
Started | 888 | 878 | 882
Vaccination 1 | 884 | 870 | 875
Vaccination 2 | 802 | 819 | 799
Vaccination 3 | 757 | 777 | 748
Completed | 722 | 733 | 717
Not Completed | 166 | 145 | 165
Not completed — Other | 9 | 8 | 6
Not completed — Medication error | 7 | 5 | 6
Not completed — Adverse Event | 12 | 5 | 6
Not completed — Protocol Violation | 12 | 19 | 16
Not completed — No longer meets eligibility criteria | 18 | 9 | 19
Not completed — Lost to Follow-up | 52 | 53 | 51
Not completed — No longer willing to participate | 52 | 38 | 54
Not completed — Randomized but not vaccinated | 4 | 8 | 7

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline | Saline+Saline+rLP2086 | Total
Number analyzed (Participants) | 888 | 878 | 882 | 2648
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.6 (0.70) | 10.6 (0.69) | 10.6 (0.67) | 10.6 (0.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 454 | 427 | 417 | 1298
  Male | 434 | 451 | 465 | 1350

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Concentrations (GMC) for Diphtheria and Tetanus Antigens
Description: Antibody GMCs of 2 antigens of diphtheria and tetanus toxoid were computed in International Units per milliliter (IU/mL) along with corresponding 2-sided 95 percent (%) confidence intervals (CIs). Here, 'number of participants analyzed' signifies participants with valid and determinate assay results for given antigen.
Time Frame: 1 Month after Vaccination 1
Population: Post vaccination 1 evaluable immunogenicity population: eligible participants randomized to Group 1 or 2, received scheduled investigational product, had pre and post vaccination blood drawn at pre-specified time points, had valid, determinate assay results for proposed analysis, received no prohibited vaccines, no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline
Number analyzed (Participants) | 778 | 780
IU/mL
  Diphtheria | 9.3 [8.67 to 9.92] | 9.8 [9.23 to 10.51]
  Tetanus | 9.4 [8.95 to 9.98] | 10.3 [9.75 to 10.85]
Statistical Analysis 1: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Diphtheria: CIs for GMC ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Diphtheria antigens); Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold and statistical inference was based on the CIs of the GMC ratios. Non-inferiority was achieved when the lower limit of the 2-sided 95% CI for the GMC ratios after vaccination 1 was greater than 0.67; GMC Ratio = 0.94, 95% CI 2-sided [0.86 to 1.03]
Statistical Analysis 2: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Tetanus: CIs for GMC ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Tetanus antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMC Ratio = 0.92, 95% CI 2-sided [0.85 to 0.99]

2. Primary Outcome: Geometric Mean Concentrations (GMC) for Acellular Pertussis Antigens
Description: Antibody GMCs of 4 acellular pertussis antigens (pertussis toxoid, pertussis filamentous hemagglutinin, pertussis pertactin and pertussis fimbrial agglutinogens types 2+3) were computed in Enzyme-linked immunosorbent assay (ELISA) units per milliliter (EU/mL) along with corresponding 2-sided 95% CIs.
Time Frame: 1 Month after Vaccination 1
Population: Post vaccination 1 evaluable immunogenicity population. Here, 'number of participants analyzed' signifies participants with valid and determinate assay results for given antigen.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline
Number analyzed (Participants) | 778 | 780
EU/mL
  Pertussis toxoid | 13.2 [12.35 to 14.14] | 14.2 [13.28 to 15.20]
  Pertussis filamentous hemagglutinin | 112.0 [106.15 to 118.14] | 122.9 [116.42 to 129.84]
  Pertussis pertactin | 202.0 [187.77 to 217.25] | 228.9 [212.72 to 246.35]
  Pertussis fimbrial agglutinogens types 2+3 | 138.1 [121.20 to 157.33] | 154.2 [135.30 to 175.79]
Statistical Analysis 1: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Pertussis toxoid: CIs for GMC ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Pertussis toxoid); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMC Ratio = 0.93, 95% CI 2-sided [0.85 to 1.02]
Statistical Analysis 2: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Pertussis filamentous hemagglutinin: CIs for GMC ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for pertussis filamentous hemagglutinin antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMC Ratio = 0.91, 95% CI 2-sided [0.84 to 0.98]
Statistical Analysis 3: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Pertussis pertactin: CIs for GMC ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for pertussis pertactin antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMC Ratio = 0.88, 95% CI 2-sided [0.80 to 0.98]
Statistical Analysis 4: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Pertussis fimbriae agglutinogens types 2 + 3: CIs for GMC ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for pertussis fimbriae agglutinogens types 2 + 3 antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; GMC Ratio = 0.90, 95% CI 2-sided [0.74 to 1.08]

3. Primary Outcome: Geometric Mean Titer (GMT) for Meningococcal Conjugate Vaccine (MCV4) Antigens
Description: Antibody GMTs of 4 MCV4 antigens (serogroup A, serogroup C, serogroup Y and serogroup W-135) were computed along with corresponding 2-sided 95% CIs.
Time Frame: 1 Month after Vaccination 1
Population: Post vaccination 1 evaluable immunogenicity population. Here, 'N' signifies participants with valid and determinate assay results for given strain for each group, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline
Number analyzed (Participants) | 779 | 781
titer
  Serogroup A (N=763, 772) | 4647.3 [4317.66 to 5002.09] | 5113.0 [4748.73 to 5505.17]
  Serogroup C (N=768, 767) | 1679.2 [1539.63 to 1831.38] | 1650.2 [1519.01 to 1792.65]
  Serogroup Y (N=771, 770) | 2212.6 [2056.08 to 2381.08] | 2244.9 [2088.70 to 2412.89]
  Serogroup W-135 (N=751, 765) | 5925.1 [5469.77 to 6418.33] | 6367.9 [5872.68 to 6904.88]
Statistical Analysis 1: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Serogroup A: CIs for GMT ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Serogroup A antigens); Test type: Non-Inferiority or Equivalence — The non-inferiority criteria margin was 1.5-fold and statistical inference was based on the CIs of the GMT ratios. Non-inferiority was achieved when the lower limit of the 2-sided 95% CI for the GMT ratios after vaccination 1 was greater than 0.67; GMT Ratio = 0.91, 95% CI 2-sided [0.82 to 1.01]
Statistical Analysis 2: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Serogroup C: CIs for GMT ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Serogroup C antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; GMT Ratio = 1.02, 95% CI 2-sided [0.90 to 1.15]
Statistical Analysis 3: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Serogroup Y: CIs for GMT ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Serogroup Y antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; GMT Ratio = 0.99, 95% CI 2-sided [0.89 to 1.09]
Statistical Analysis 4: Comparison: MCV4+Tdap+rLP2086 vs MCV4+Tdap+Saline; Serogroup W-135: CIs for GMT ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for Serogroup W-135 antigens); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; GMT Ratio = 0.93, 95% CI 2-sided [0.83 to 1.04]

4. Primary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) GMTs of PMB80 [A22] and PMB2948 [B24] 1 Month After Vaccination 3
Description: Antibody hSBA GMTs of primary strain PMB80 [A22] and PMB2948 [B24] were computed along with corresponding 2-sided 95% CIs. hSBA titers from the 2 primary strains were logarithmically transformed for analysis. Here, 'number of participants analyzed' signifies evaluable immunogenicity population and 'N' signifies participants with valid and determinate assay results for given strain for each group, respectively.
Time Frame: 1 Month after Vaccination 3
Population: Post vaccination 3 evaluable immunogenicity population: eligible participants randomized to Group 1 or 3, received scheduled investigational product, had pre and post vaccination blood drawn at pre-specified time points, had valid, determinate assay results for proposed analysis, received no prohibited vaccines, no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MCV4+Tdap+rLP2086 | Saline+Saline+rLP2086
Number analyzed (Participants) | 683 | 679
titer
  PMB80 [A22] (N=679, 674) | 45.9 [42.74 to 49.35] | 49.7 [46.43 to 53.30]
  PMB2948 [B24] (N=670, 656) | 24.8 [23.11 to 26.58] | 27.4 [25.58 to 29.41]
Statistical Analysis 1: Comparison: MCV4+Tdap+rLP2086 vs Saline+Saline+rLP2086; PMB80 [A22]: CIs for GMT ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for hSBA strain titers); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; GMT Ratio = 0.92, 95% CI 2-sided [0.84 to 1.02]
Statistical Analysis 2: Comparison: MCV4+Tdap+rLP2086 vs Saline+Saline+rLP2086; PMB2948 [B24]: CIs for GMT ratio were back transformations of a confidence interval based on the Student t distribution for the mean difference of the logarithms of the measures (Group 1 - Group 2 for hSBA strain titers); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; GMT Ratio = 0.90, 95% CI 2-sided [0.82 to 1.00]

5. Secondary Outcome: Percentage of Participants With Seroresponse for Tetanus, Diphtheria and Acellular Pertussis (Tdap) and Meningococcal Conjugate Vaccine (MCV4) Antigens
Description: Seroconversion rate for Tdap antigens was defined as greater than or equal to (>=) 4-, 2-fold rise in antibody concentration, if prevaccination antibody concentration was less than or equal to (<=), greater than (>) cutoff value, respectively. For MCV4 antigens >=4-fold rise on serum bactericidal assay using rabbit complement (rSBA) titers if baseline value >= lower limit of quantitation (LLOQ), postdose rSBA titers >=2×LLOQ if baseline value was less than (<) LLOQ. Cutoff value =0.1 IU/mL for diphtheria and tetanus, 0.9,2.9,3.0,10.6 EU/mL for pertussis toxoid, filamentous hemagglutinin, pertactin, fimbriae agglutinogens types 2 + 3, respectively.
Time Frame: 1 Month after Vaccination 1
Population: Post vaccination 1 evaluable immunogenicity population. Here, 'number of participants analyzed' signifies participants with valid, determinate assay results for given antigen at specified time point and baseline. 'N' signifies number of participants with seroresponse.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline
Number analyzed (Participants) | 779 | 781
percentage of participants
  Diphtheria (N=774, 780) | 98.6 [97.5 to 99.3] | 98.3 [97.2 to 99.1]
  Tetanus (N=774, 780) | 97.7 [96.3 to 98.6] | 97.4 [96.1 to 98.4]
  Pertussis toxoid (N=774, 780) | 68.1 [64.7 to 71.4] | 72.7 [69.4 to 75.8]
  Pertussis filamentous hemagglutinin (N=774, 780) | 85.3 [82.6 to 87.7] | 89.2 [86.8 to 91.3]
  Pertussis pertactin (N=774, 780) | 96.0 [94.4 to 97.3] | 96.2 [94.6 to 97.4]
  Pertussis fimbriae AG types 2+3 (N=774, 780) | 79.5 [76.4 to 82.3] | 81.9 [79.0 to 84.6]
  Serogroup A (N=712, 736) | 85.4 [82.6 to 87.9] | 88.6 [86.1 to 90.8]
  Serogroup C (N=738, 742) | 89.3 [86.8 to 91.4] | 88.9 [86.5 to 91.1]
  Serogroup Y (N=754, 753) | 90.5 [88.1 to 92.5] | 93.6 [91.6 to 95.3]
  Serogroup W-135 (N=729, 752) | 97.1 [95.6 to 98.2] | 97.2 [95.8 to 98.3]

6. Secondary Outcome: Percentage of Participants Achieving Predefined Antibody Level for Diphtheria and Tetanus Antigens
Description: Participants with antibody concentration level of greater than or equal to 1.0 IU/mL for diphtheria and tetanus antigens were computed along with corresponding 2-sided 95% CIs.
Time Frame: 1 Month after Vaccination 1
Population: Post vaccination 1 evaluable immunogenicity population. Here, 'number of participants analyzed' signifies participants with valid, determinate assay results for given antigen.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline
Number analyzed (Participants) | 778 | 780
percentage of participants
  Tetanus | 99.1 [98.2 to 99.6] | 99.0 [98.0 to 99.6]
  Diphtheria | 98.1 [96.8 to 98.9] | 99.0 [98.0 to 99.6]

7. Secondary Outcome: Serum Bactericidal Assay Using Human Complement (hSBA) GMTs of PMB80 [A22] and PMB2948 [B24] Before Vaccination 1 and 1 Month After Vaccination 2
Description: Antibody hSBA of primary strain PMB80 [A22] and PMB2948 [B24] were computed along with corresponding 2-sided 95% CIs. hSBA titers from the 2 primary strains were logarithmically transformed for analysis.
Time Frame: Before Vaccination 1, 1 Month after Vaccination (Vac) 2
Population: Post vaccination 3 evaluable immunogenicity population. Here, 'number of participants analyzed' signifies evaluable immunogenicity population and 'N' signifies participants with valid and determinate assay results for given strain for each group, respectively.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | MCV4+Tdap+rLP2086 | Saline+Saline+rLP2086
Number analyzed (Participants) | 683 | 679
titer
  Before Vaccination 1: PMB80 [A22] (N=677, 677) | 8.5 [8.28 to 8.64] | 8.6 [8.39 to 8.84]
  Before Vaccination 1: PMB2948 [B24] (N=677, 676) | 4.1 [4.04 to 4.19] | 4.2 [4.10 to 4.27]
  1 Month after Vac 2: PMB80 [A22] (N=669, 665) | 23.7 [22.10 to 25.40] | 23.8 [22.14 to 25.54]
  1 Month after Vac 2: PMB2948 [B24] (N=656, 650) | 12.0 [11.12 to 12.99] | 13.0 [12.03 to 14.13]

8. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer >= Lower Limit of Quantitation (LLOQ)
Description: Percentage of participants achieving hSBA titer >= LLOQ were computed along with corresponding 2-sided 95% CIs. LLOQ was 1:16 for PMB80 [A22] and 1:8 for PMB2948 [B24].
Time Frame: Before Vaccination 1, 1 Month after Vaccination (Vac) 2, 3
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MCV4+Tdap+rLP2086 | Saline+Saline+rLP2086
Number analyzed (Participants) | 683 | 679
percentage of participants
  Before Vaccination 1: PMB80[A22] 1:16 (N=677, 677) | 4.4 [3.0 to 6.3] | 5.6 [4.0 to 7.6]
  1 month after Vac 2: PMB80[A22] 1:16 (N= 669, 665) | 68.0 [64.3 to 71.5] | 68.0 [64.3 to 71.5]
  1 month after Vac 3: PMB80 [A22] 1:16 (N=679, 674) | 87.5 [84.8 to 89.9] | 91.4 [89.0 to 93.4]
  Before Vaccination 1: PMB2948[B24] 1:8 (N=677,676) | 1.6 [0.8 to 2.9] | 3.4 [2.2 to 5.1]
  1 month after Vac 2: PMB2948[B24] 1:8 (N=656, 650) | 62.3 [58.5 to 66.1] | 66.0 [62.2 to 69.6]
  1 month after Vac 3: PMB2948[B24] 1:8 (N=670, 656) | 90.0 [87.5 to 92.2] | 92.7 [90.4 to 94.6]

9. Secondary Outcome: Percentage of Participants With Serum Bactericidal Assay Using Human Complement (hSBA) Titer >= Prespecified Titer Level
Description: Antibody hSBA of primary strain PMB80 [A22] and PMB2948 [B24] with hSBA titers >=1:4, >=1:8, >=1:16, >=1:32, >=1:64, and >=1:128 were computed along with corresponding 2-sided 95% CIs.
Time Frame: Before Vaccination 1, 1 Month after Vaccination (Vac) 2, 3
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MCV4+Tdap+rLP2086 | Saline+Saline+rLP2086
Number analyzed (Participants) | 683 | 679
percentage of participants
  Before Vaccination 1: PMB80[A22] 1:4 (N=677,677) | 6.9 [5.1 to 9.1] | 7.5 [5.7 to 9.8]
  1 month after Vac 2: PMB80[A22] 1:4 (N=669, 665) | 68.2 [64.5 to 71.7] | 68.6 [64.9 to 72.1]
  1 month after Vac 3: PMB80[A22] 1:4 (N=679, 674) | 87.8 [85.1 to 90.1] | 91.7 [89.3 to 93.7]
  Before Vaccination 1: PMB80[A22] 1:8 (N=677, 677) | 5.0 [3.5 to 6.9] | 6.4 [4.6 to 8.5]
  1 month after Vac 2: PMB80[A22] 1:8 (N=669, 665) | 68.2 [64.5 to 71.7] | 68.1 [64.4 to 71.7]
  1 month after Vac 3: PMB80[A22] 1:8 (N=679, 674) | 87.6 [84.9 to 90.0] | 91.5 [89.2 to 93.5]
  Before Vaccination 1: PMB80[A22] 1:32 (N=677, 677) | 2.7 [1.6 to 4.2] | 3.2 [2.0 to 4.9]
  1 month after Vac 2: PMB80[A22] 1:32 (N=669, 665) | 55.0 [51.1 to 58.8] | 54.4 [50.6 to 58.3]
  1 month after Vac 3: PMB80[A22] 1:32 (N=679, 674) | 81.3 [78.2 to 84.2] | 84.7 [81.8 to 87.4]
  Before Vaccination 1: PMB80[A22] 1:64 (N=677,677) | 0.7 [0.2 to 1.7] | 1.0 [0.4 to 2.1]
  1 month after Vac 2: PMB80[A22] 1:64 (N= 669, 665) | 25.6 [22.3 to 29.0] | 25.0 [21.7 to 28.4]
  1 month after Vac 3: PMB80[A22] 1:64 (N=679, 674) | 52.7 [48.9 to 56.5] | 55.6 [51.8 to 59.4]
  Before Vaccination 1: PMB80[A22] 1:128 (N=677,677) | 0.1 [0.0 to 0.8] | 0.4 [0.1 to 1.3]
  1 month after Vac 2: PMB80[A22] 1:128 (N=669, 665) | 6.9 [5.1 to 9.1] | 7.5 [5.6 to 9.8]
  1 month after Vac 3: PMB80[A22] 1:128 (N=679, 674) | 23.6 [20.4 to 26.9] | 23.3 [20.2 to 26.7]
  Before Vaccination 1: PMB2948[B24] 1:4 (N=677,676) | 2.1 [1.1 to 3.4] | 3.7 [2.4 to 5.4]
  1 month after Vac 2: PMB2948[B24] 1:4 (N=656, 650) | 64.8 [61.0 to 68.4] | 68.2 [64.4 to 71.7]
  1 month after Vac 3: PMB2948[B24] 1:4 (N=670, 656) | 90.7 [88.3 to 92.8] | 93.1 [90.9 to 95.0]
  Before Vaccination 1: PMB2948[B24] 1:16(N=677,676) | 1.5 [0.7 to 2.7] | 2.1 [1.1 to 3.5]
  1 month after Vac 2: PMB2948[B24] 1:16(N=656,650) | 57.6 [53.7 to 61.4] | 60.3 [56.4 to 64.1]
  1 month after Vac 3: PMB2948[B24] 1:16(N=670,656) | 86.7 [83.9 to 89.2] | 88.9 [86.2 to 91.2]
  Before Vaccination 1: PMB2948[B24] 1:32(N=677,676) | 0.4 [0.1 to 1.3] | 0.6 [0.2 to 1.5]
  1 month after Vac 2: PMB2948[B24] 1:32(N=656,650) | 26.2 [22.9 to 29.8] | 28.2 [24.7 to 31.8]
  1 month after Vac 3: PMB2948[B24] 1:32(N=670, 656) | 55.1 [51.2 to 58.9] | 60.7 [56.8 to 64.4]
  Before Vaccination 1:PMB2948[B24] 1:64(N= 677,676) | 0.4 [0.1 to 1.3] | 0.3 [0.0 to 1.1]
  1 month after Vac 2: PMB2948[B24] 1:64 (N=656,650) | 8.7 [6.6 to 11.1] | 10.3 [8.1 to 12.9]
  1 month after Vac 3: PMB2948[B24] 1:64 (N=670,656) | 22.5 [19.4 to 25.9] | 24.1 [20.9 to 27.5]
  Before Vaccination 1:PMB2948[B24] 1:128(N=677,676) | 0.1 [0.0 to 0.8] | 0.1 [0.0 to 0.8]
  1 month after Vac 2: PMB2948[B24] 1:128(N=656,650) | 2.4 [1.4 to 3.9] | 3.4 [2.1 to 5.1]
  1 month after Vac 3: PMB2948[B24] 1:128(N=670,656) | 6.6 [4.8 to 8.7] | 7.8 [5.8 to 10.1]

10. Other Pre Specified Outcome: Immunogloblulin G (IgG) Measured by GMC
Description: IgG GMCs of 4 MCV4 antigens (serogroup A, serogroup C, serogroup Y and serogroup W-135) of participants were computed along with corresponding 2-sided 95% CIs. CIs were back transformations of confidence levels based on Student t distribution for mean logarithm of titers.
Time Frame: Before Vaccination 1, 1 Month after Vaccination 1
Population: Post vaccination 1 evaluable immunogenicity population.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter (mcg/mL)
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline
Number analyzed (Participants) | 779 | 781
microgram per milliliter (mcg/mL)
  Before Vaccination 1: Serogroup A | 0.17 [0.16 to 0.19] | 0.15 [0.14 to 0.17]
  1 Month after Vaccination 1: Serogroup A | 11.42 [10.30 to 12.65] | 11.38 [10.21 to 12.67]
  Before Vaccination 1: Serogroup C | 0.11 [0.10 to 0.12] | 0.11 [0.10 to 0.12]
  1 Month after Vaccination 1: Serogroup C | 5.59 [4.90 to 6.39] | 5.47 [4.79 to 6.23]
  Before Vaccination 1: Serogroup Y | 0.14 [0.13 to 0.14] | 0.13 [0.13 to 0.14]
  1 Month after Vaccination 1: Serogroup Y | 2.49 [2.22 to 2.79] | 2.14 [1.92 to 2.39]
  Before Vaccination 1: Serogroup W-135 | 0.13 [0.13 to 0.14] | 0.13 [0.13 to 0.14]
  1 Month after Vaccination 1: Serogroup W-135 | 1.79 [1.59 to 2.01] | 1.84 [1.62 to 2.09]

11. Other Pre Specified Outcome: Percentage of Participants Achieving at Least 4-Fold Increase in Serum Bactericidal Assay Using Human Complement (hSBA) Titer Level
Time Frame: 1 Month after Vaccination (Vac) 2, 3
Population: Post vaccination 3 evaluable immunogenicity population. Here, 'number of participants analyzed' signifies evaluable immunogenicity population and 'N' signifies participants with valid and determinate hSBA titers for the given strain at both the specified time point and baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MCV4+Tdap+rLP2086 | Saline+Saline+rLP2086
Number analyzed (Participants) | 683 | 679
percentage of participants
  1 month after Vac 2 : PMB80 [A22] (N=663, 663) | 64.3 [60.5 to 67.9] | 63.7 [59.9 to 67.3]
  1 month after Vac 3 : PMB80 [A22] (N=673, 672) | 84.0 [81.0 to 86.6] | 88.7 [86.0 to 91.0]
  1 month after Vac 2 : PMB2948 [B24] (N=650, 647) | 56.3 [52.4 to 60.2] | 58.4 [54.5 to 62.3]
  1 month after Vac 3 : PMB2948 [B24] (N=664, 653) | 85.7 [82.8 to 88.3] | 87.7 [85.0 to 90.2]

12. Other Pre Specified Outcome: Percentage of Participants With at Least One Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship.
Time Frame: Vaccination phase (baseline up to 1 month after Vaccination 3); Follow-up phase (from 1 month up to 6 months after Vaccination 3)
Population: Safety population included all participants who received at least 1 dose of the investigational product and had safety information available. 'N' signifies participants evaluable for this measure during specified time period.
Measure: Number; unit: percentage of participants
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline | Saline+Saline+rLP2086
Number analyzed (Participants) | 883 | 870 | 875
percentage of participants
  Vaccination phase: Adverse Events (N=883,870,875) | 42.9 | 42.6 | 46.2
  Follow-up phase: Adverse Events (N=777,776,771) | 1.0 | 0.5 | 1.3

ADVERSE EVENTS:
Time Frame: AEs: recorded from signing of informed consent form (ICF) to completion of study. SAEs: recorded from signing of ICF to 196 days of follow up period. Participant recorded pre--specified AEs in electronic diary (up to 7 days after vaccination)
Description: SAEs and AEs were grouped by system organ class and preferred term. AEs included AEs collected in the electronic diary (local and systemic reactions; systematic assessment) and AEs collected on the case report form at each visit (nonsystematic assessment).
Arm/Group | MCV4+Tdap+rLP2086 | MCV4+Tdap+Saline | Saline+Saline+rLP2086
Serious Adverse Events (participants affected / at risk) | 15/883 | 9/870 | 11/875
Other Adverse Events (participants affected / at risk) | 277/883 | 260/870 | 292/875
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCV4+Tdap+rLP2086 (N=883) | MCV4+Tdap+Saline (N=870) | Saline+Saline+rLP2086 (N=875)
Adrenogenital syndrome (Congenital, familial and genetic disorders) | 1 | 0 | 0
Congenital spinal cord anomaly (Congenital, familial and genetic disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0 | 1
Bone abscess (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Epiphyseal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 1
Dural arteriovenous fistula (Nervous system disorders) | 1 | 0 | 0
Hemiplegic migraine (Nervous system disorders) | 0 | 0 | 1
Migraine (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Affective disorder (Psychiatric disorders) | 1 | 1 | 0
Depression suicidal (Psychiatric disorders) | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 0 | 1
Encopresis (Psychiatric disorders) | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0
Psychogenic seizure (Psychiatric disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MCV4+Tdap+rLP2086 (N=883) | MCV4+Tdap+Saline (N=870) | Saline+Saline+rLP2086 (N=875)
Vomiting (Gastrointestinal disorders) | 18 | 21 | 19
Nausea (Gastrointestinal disorders) | 10 | 9 | 14
Abdominal pain (Gastrointestinal disorders) | 2 | 7 | 10
Injection site pain (General disorders) | 19 | 21 | 15
Pyrexia (General disorders) | 20 | 14 | 17
Upper respiratory tract infection (Infections and infestations) | 47 | 61 | 70
Pharyngitis (Infections and infestations) | 38 | 27 | 28
Pharyngitis streptococcal (Infections and infestations) | 23 | 20 | 30
Nasopharyngitis (Infections and infestations) | 22 | 19 | 16
Gastroenteritis viral (Infections and infestations) | 15 | 15 | 25
Gastroenteritis (Infections and infestations) | 15 | 20 | 16
Sinusitis (Infections and infestations) | 18 | 13 | 17
Otitis media (Infections and infestations) | 17 | 11 | 14
Bronchitis (Infections and infestations) | 5 | 6 | 15
Viral infection (Infections and infestations) | 4 | 7 | 12
Conjunctivitis (Infections and infestations) | 9 | 6 | 3
Otitis externa (Infections and infestations) | 17 | 11 | 14
Fall (Injury, poisoning and procedural complications) | 12 | 13 | 16
Ligament sprain (Injury, poisoning and procedural complications) | 12 | 12 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 4 | 8
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 | 2 | 3
Headache (Nervous system disorders) | 24 | 29 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 20 | 31
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 17 | 13 | 23
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 11
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 10
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 9
Dermatitis contact (Skin and subcutaneous tissue disorders) | 11 | 1 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other